CLINICAL TRIAL: NCT06421246
Title: Physical Activity in Geriatric Patients Before and After the Introduction of a Staff-facing Real-time Activity Screen and Validation of the Danish Version of the Acute Care Mobility Assessment - a Hybrid Implementation and Effectiveness Study in Two Patient Cohorts
Brief Title: Implementation and Evaluation of Real Time Monitoring of Physical Activity in Geriatric Patients - a Hybrid Implementation and Effectiveness Study in Two Patient Cohorts
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mette Merete Pedersen, Senior Researcher, Copenhagen University Hospital, Hvidovre
Other Study IDs: F-24023831
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Disease; Old Age
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Activity monitoring and validity of the Danish Version of the Acute Care Mobility Assessement: 24- hour activity will be assessed by SENS motion acitivity monitors before (Cohort 1) and after the introduction (Cohort 2) of a screen-solution with staff-facing real time activity data and investigation of the implementation process and outcomes. Furthermore, the Acute Care mobility assessment will be validated by cognitive debriefing interviews in 5-10 patients in Cohort 1.
  Interventions: Behavioral: Staff-facing screen

INTERVENTIONS:
Behavioral: Staff-facing screen — Activity will be monitored before and after the introduction of a staff-facing screen

SUMMARY:
The study aim to assess 24-hour activity during hospitalization in older adults admitted to a geriatric ward and to validate the Danish version of the Acute Care Mobility Assessment.

In a follow-up study, we will implement and evaluate a staff-facing activity screen showing real-time physical activity in the geriatric ward with a focus on changes in staff culture (awareness and actions) and basis for data-driven discussions about physical activity during hospitalization inspired by Making Every Contact Count. Also, we will reassess in-hospital physical activity in older adults admitted to the geriatric ward.

DETAILED DESCRIPTION:
The study uses a Hybrid Type I design in which both the implementation of a staff-facing screen and the effectiveness on physical activity will be evaluated. The study is conducted in two phases.

Phase one is an observational cohort study. During 6 weeks, 24-hour activity will be assessed in all patients (65+) admitted to a geriatric ward in Denmark, who are able to walk and to provide informed consent (or vicarious consent). Activity will be measured for a maximum of 7 days. Demographic characteristics will be collected (sex, age, place of residence, comorbidities, admission diagnosis, civil status, frailty), and the patients will be asked about their: daily activities, walking ability, life space activity, present activity, use of walking aids, and falls. On inclusion, the patients will be assessed for their basic mobility, cognition, gait speed, and their level of mobility. The Acute Care Mobility Assessment will be validated on the initial 5-10 patients via cognitive debriefing interviews (May-July 2024). In the same period, an ethnographic field study will be conducted with focus on physical activity followed by semi-structured interviews (N=17) with managers and health care professionals.

In the follow-up study, we will assess in-hospital physical activity over a 6-week period after introducing a staff-facing activity screen, showing real-time activity and to investigate whether the activity screen increases physical activity among hospitalized geriatric patients. 24-hours physical activity will be re-quantified using SENS motion ®, sensor technology. The study design will otherwise follow the same approach as the initial study, including the use of the same outcome measures. In the same period, we will repeat the ethnographic field study and interviews regarding focus on physical activity and implementation of the activity screen with managers and health care professionals inspired by Making Every Contact Count. The Consolidated Framework for Implementation Research (CFIR) will be used as Framework, and focus will be on adoption and adaptation.

The study meets the guidelines of the Declaration of Helsinki and is approved by the Research Ethics Committee (F-24023831).

ELIGIBILITY:
Inclusion Criteria:

* 65 years
* no delirium
* ability to ambulate

Exclusion Criteria:

* in isolation
* teminally ill
* Expected to be discharged within 24-hours from inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults admitted to a geriatric ward at Copenhagen University Hospital, Hvidovre
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily steps | 7 days
  Number of daily steps taken and the distribution over the entire hospitalization, assessed by a SENS motion accelerometer from inclusion and throughout hospitalization.

SECONDARY OUTCOMES:
Self-reported mobility | Days 2, 4 and 6 after inclusion
  Self-reported mobility by the Acute Care Mobility Assessment. A score of 0-12 can be obtained, with 0 reflecting poor mobility and 12 reflecting a high level of mobility.
Life Space mobility | At inclusion, 4 weeks post discharge
  By the Life Space Assessment-DK, which measure mobility and level of dependence in mobility. A score of 0-120 can be obtained, with 0 reflecting poor mobility and 120 reflecting high mobility.
Self-reported pre-admission (2 weeks prior to admission) and post discharge mobility | At inclusion and 1 week after discharge
  By the New Mobility Score, which assesses the ability to walk indoors and outdoors and the ability to go shopping. A score from 0-9 can be obtained, with 0 reflecting low mobility and 9 reflecting high mobility.
Frailty | At inclusion
  By the Clinical Frailty Scale, which is a clinical evaluation of the degree of frailty of a person. It is scored by health care professionals on a scale from 1 (very fit) to 9 (terminally ill)
Cognitive status | At inclusion
  By the Orientation Memory Concentration Test, which is a screening of cognitive function. A score from 0 to 28 i obtained with lower scores reflecting poorer cognition (0-7: highly impaired; 8-17 points: moderately imparied; 18-24 points: mildly impaired; 25-28 points: no or insignificatn impairment).
Activities of daily living | At inclusion and 1 week after discharge
  By the Katz index, which assesses independence in 6 Activities of Daily Living on a scale from 0 to 6 with 0 reflecting dependence in all activities and 6 reflecting independence in all activities.
Basic mobility | Days 2, 4 and 6 after inclusion
  By the The Cummulated Ambulation Score, which assessed the ability of a person to get in an out of bed, sit to stand from a chair and walk. It is scored from 0 to 6 with 0 reflecting inability to perform the 3 activities and a score of 6 refelcting independence in the three activities.
Highest level of mobility | At inclusion
  By the Johns Hopkins Higest Level of Mobility Scale which evaluates a patient's level of mobiltiy on a 1 (lying) to 8 (waling more than 250 feet) point scale
Gait speed | At inclusion
  By the 4 meter habitual gait speed test. It assesses the patient's habitual gait speed on a 4-meter course. The test is scored in m/s.
Uptime | 7 days
  Daily time spent in uptime and the distribution over the entire hospitalization, assessed by a SENS motion accelerometer from inclusion and throughout hospitalization.
Daily walking | 7 days
  Daily time spent walking and the distribution over the entire hospitalization, assessed by a SENS motion accelerometer from inclusion and throughout hospitalization.
Daily standing | 7 days
  Daily time spent walking assessed by a SENS motion accelerometer from inclusion and throughout hospitalization.
Daily lying/sitting | 7 days
  Daily time spent sitting/lying and the distribution over the entire hospitalization, assessed by a SENS motion accelerometer from inclusion and throughout hospitalization.
Readmission | 3 months after discharge
  Number of readmission with three months after discharge
Falls | 1 month after discharge
  Number of falls within the first month after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansen LK, Larsen TS, Kirk JW, Pedersen BS, Nielsen BR, Kallemose T, Bandholm T, Pedersen MM. Exploring in-hospital mobility practices for geriatric patients: insights from a mixed-method study. BMC Geriatr. 2025 May 13;25(1):330. doi: 10.1186/s12877-025-05976-9. PMID 40361036